CLINICAL TRIAL: NCT06263322
Title: ROAMM-EHR: Pilot Trial of a Real-Time Symptom Surveillance System for Post-Discharge Surgical Patients
Brief Title: The ROAMM-EHR Study
Acronym: ROAMM-EHR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB202200419; R21AG073769 (NIH)
Record Dates: First submitted 2024-02-09; First posted 2024-02-16 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: Parallel Randomized Clinical trial. Comparison study to test the feasibility of patient generated health data compared to standard of care post-surgical observation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants are masked to whether their PGHD are being sent to their care provider. Care providers are masked to who receives standard of care. Investigators (except for one who will be the point person for randomization) will be masked to intervention assignments. Staff assessors will be masked to whether PGHD are being sent to their care provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROAMM-EHR (Experimental): Patients will wear a smartwatch equipped with a smartwatch app before their surgery and for approximately a month after the surgery. Patients will be asked to wear the watch every day when awake. When wearing the smartwatch, patients will be asked questions about their symptoms following surgery and data will be sent to providers electronically and displayed in their EHR portal. Healthcare Providers will use this information along with patient medical history to decide on the next course of action. The study does not provide specific instructions about how to care for the patient. Those decisions are made by the provider team and their clinical judgement.
  Interventions: Behavioral: Actionable remotely generated health data
- Active Comparison (Active Comparator): The active comparison patients will wear and respond to questions on the smartwatch. However, the information will not be viewable by their doctor and medical team. All standard of care procedures will remain.
  Interventions: Behavioral: Non-Actionable remotely generated health data

INTERVENTIONS:
Behavioral: Actionable remotely generated health data — Remotely captured, patient generated health data will be used to inform provider care following re-vascular surgery in patients with chronic limb threatening ischemia
  Arms: ROAMM-EHR
Behavioral: Non-Actionable remotely generated health data — Remotely captured, patient generated health data is captured, but will not be used to inform provider care following re-vascular surgery in patients with chronic limb threatening ischemia
  Arms: Active Comparison

SUMMARY:
In recent years, mobile health (mHealth) apps have promised improved monitoring of health conditions to improve clinical outcomes. The objective of this study is to conduct a pilot randomized clinical trial (RCT) to evaluate the impact of using remotely collected patient generated health data (PGHD) from older patients undergoing bypass surgery due to chronic limb threatening ischemia. The hypothesis is that integrating PGHD with an EHR system will help providers manage post-surgical symptoms and thus improve post-operative mobility and quality of life health outcomes.

DETAILED DESCRIPTION:
This pilot study aims to evaluate the feasibility of collecting patient generated health data (PGHD) remotely for aiding care management of patients with chronic limb threatening ischemia following vascular bypass or revascularization. DRemote data collected from a publicly available smartwatch will be displayed on an EHR interface for providers to view PGHD. The test of feasibility entails multiple components that include implementing a provider interface for viewing and acting on PGHD, establishing safety, ensuring quality assurance (e.g. quality of remote data collection), successful recruitment and retention of participants, and sufficient remote response rates from patients.

ELIGIBILITY:
Inclusion Criteria:

* age >= 60; Patients with chronic limb threatening ischemia who are undergoing re-vascular surgery [endovascular or open re-vascularization (bypass)].

Exclusion Criteria:

* High risk of post-surgical amputation based on study physician judgement, non-english speaker, diagnosis of an age-related dementia (e.g. Alzheimer's Disease); unable to communicate because of severe hearing loss; uncorrectable vision impairment that compromises clinical assessments or would cause a safety concern, other significant co-morbid disease that in the opinion of the investigators and study physician would impair the ability to participate in the study or be a safety concern

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2026-10-17 (Estimated); Study Completion 2026-10-17 (Estimated)

PRIMARY OUTCOMES:
6-min walk distance | Baseline and approximately 30 days post-surgery
  Patients are asked to complete as much distance as possible over a standardized course

SECONDARY OUTCOMES:
self-reported quality of life | Baseline and approximately 30 days post-surgery
  Outcome will be assessed as the summary score on the Medical Outcomes Study 36-Item Short Form (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Manini, PhD, Principal Investigator — University of Florida
Locations (1):
- Institute of Aging, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study that tests feasibility. Collection of data for definitive testing purposes is not appropriate at this stage. If the study tests as feasible we will pursue data sharing under policies set forth by the local institution, privacy office and regulatory authorities. We will also follow any journal requirements for posting deidentified data.